CLINICAL TRIAL: NCT00374387
Title: Psychosocial and Physiological Mechanisms in the Effect of Hormonal Contraception on the Female Sexual Desire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Petra De Sutter, University Hospital Ghent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006/309
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Healthy women
MeSH Terms: interventions — NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nuvaring
Drug: low-dose combination pill
Drug: minipill

SUMMARY:
75 heterosexual women are asked to use 3 different types of contraception (Nuvaring, low-dose combination pill, minipill), each during 3 months. On a monthly basis, questionnaires are filled out about sexual desire and psychosocial, relational en sexual parameters. Also the sexual desire of the partner is questioned. On a three-monthly basis, blood samples are drawn to determine changes in hormonal parameters (one sample per product period).

75 lesbian women are doing the same trial, but during an extra 3 months period, they are asked to have their natural menstrual cyclus as a control condition. Blood samples during these extra months will be drawn at the third or fourth day after start of the menses.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual or lesbian women
* Aged between 18 and 45 years
* Stable monogameous relationship
* Normal menstrual cyclus

Exclusion Criteria:

* Polycystic ovarial syndrome
* Normal exclusion criteria for the use of contraception
* Use of medication known to influence sexual desire and/or androgen levels
* Women who wants to become pregnant, are pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Parameters about sexual desire and psychosocial, relational en sexual parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Petra De Sutter, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be